CLINICAL TRIAL: NCT05285540
Title: A Phase 1a, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of DT-216 in Adult Patients With Friedreich Ataxia
Brief Title: Study to Evaluate DT-216 in Adult Patients With Friedreich Ataxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Design Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTX-216-101
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Dose: DT-216 (Experimental): DT-216 will be administered once
  Interventions: Drug: DT-216
- Single Dose: DT-216 matching placebo (Experimental): Placebo will be administered once
  Interventions: Drug: DT-216 matching Placebo

INTERVENTIONS:
Drug: DT-216 — DT-216 will be administered by intravenous (IV) injection
  Arms: Single Dose: DT-216
Drug: DT-216 matching Placebo — Placebo will be administered by intravenous (IV) injection
  Arms: Single Dose: DT-216 matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic effects of intravenous DT-216 in adult patients with Friedreich Ataxia. This single ascending dose study is randomized, double-blind, placebo-controlled.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Friedreich Ataxia with homozygous GAA repeat expansions
* Body mass index (BMI) between 17 and 32 kg/m2
* Stage 5.5 or less on the Functional Staging for Ataxia (FSA)

Exclusion Criteria:

* Has any concomitant medical condition that in the opinion of the investigator, puts the participant at risk or precludes participant from completing the study
* Has clinically significant abnormal laboratory results
* Has significant cardiac disease
* Received an investigational drug within 3 months of screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment adverse events (TEAEs) | Up to approximately 30 days
  Frequency of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of DT-216 | Up to approximately 30 days
  Maximum Plasma Concentration (Cmax) of DT-216
Time to Maximum Plasma Concentration (Tmax) of DT-216 | Up to approximately 30 days
  Time to Maximum Plasma Concentration (Tmax) of DT-216
Area Under the Concentration-time Curve (AUC) of DT-216 | Up to approximately 30 days
  Area Under the Concentration-time Curve (AUC) of DT-216

OTHER OUTCOMES:
Frataxin expression | Up to approximately 30 days
  Frataxin mRNA and protein expression measured in peripheral blood monocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinilabs, Eatontown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No